CLINICAL TRIAL: NCT06043232
Title: The Role and Mechanism of MMR/MSI Phenotypes in Evaluating Vaccine Benefit in Glioblastoma
Brief Title: MMR/MSI Phenotypes in Prediction of Tumor Vaccine Benefit for Gliomas
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Yao, MD, Professor, Huashan Hospital
Other Study IDs: KY2023-520
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Glioma
Keywords: Glioblastoma multiforme; DC vaccine; Mismatch repair; Microsatellite instability; Biomarker
MeSH Terms: conditions — Glioma; Glioblastoma; Microsatellite Instability | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- glioma patients with routine surgery: surgery
- glioma patients with DC vaccine: surgery and DC vaccine
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — DC vaccine produced by the Team
  Groups: glioma patients with DC vaccine

SUMMARY:
Glioblastoma (GBM) is the most malignant primary intracranial tumor with a median survival of about 18 months, and new therapies are urgently needed. Tumor vaccines has been shown to improve survival of GBM, but not all patients can benefit from vaccine treatment and biomarkers are urgently needed. Deletion of mismatch repair (MMR) protein and microsatellite instability (MSI) state are important features in the biological evolution of GBM, and may be used as markers for tumor vaccine. Therefore, this project will collect samples from GBM patients before and after vaccine treatment respectively, and evaluate the role of MMR/MSI gene phenotype in predicting vaccine efficacy and the potential molecular mechanism. Moreover, MMR/MSI phenotypes will be assessed by deep-learning and radiomics using images to establish noninvasive markers for vaccine.

ELIGIBILITY:
Inclusion Criteria:

The patients with glioma in the Department of Neurosurgery of Huashan Hospital Affiliated to Fudan University who meet the following three conditions can be enrolled

1. They were 18-80 years old, male and female;
2. The pathological results of frozen section during operation were gliomas (20 cases of who grade II, II and IV, respectively);
3. Tissue (6 mm * 6 mm) can be used for cell sorting on the basis of not affecting clinical routine diagnosis;
4. Sign informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will not be included in this study:

1. Participants in other clinical trials;
2. Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioma surgery at Huashan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics | 36 months
  The issues collected will be used for transcriptome sequencing to measure gene expression level.
Immunomics | 36 months
  The issues collected will be used for TCR/BCR sequencing to measure clonality of lymphocytes
Proteomics | 36 months
  The issues collected will be used for TCR/BCR sequencing to measure gene expression level in protein
Radiomics | 36 months
  The features from images will be extracted using algorithm of Deep-learning or Radiomics
IHC analysis | 36 months
  Different expression level of proteins (CD3,CD8,B7-H4, MMR proteins) in Gliomas with different grades and molecular subgroups (300 cases) will be measured using immunohistochemical.
Genomics | 36 months
  The issues collected will be used for whole genome sequencing or whole exome sequencing to measure gene mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital，Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No